CLINICAL TRIAL: NCT01563783
Title: The Trust (Treatment Results of Uterine Sparing Technologies) Study
Brief Title: Post Market TRUST Study
Acronym: TRUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acessa Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-00-0015
Record Dates: First submitted 2012-03-22; First posted 2012-03-27 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Uterine Fibroids
Keywords: Fibroids; Myomas; leiomyomata; menorrhagia; Acessa Procedure; Radiofrequency Ablation; RFA
MeSH Terms: conditions — Leiomyoma; Myoma; Menorrhagia | interventions — Uterine Myomectomy; Uterine Artery Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Woman Suitable for Myomectomy or GFA (Active Comparator): This group will consist of women who desire uterine preservation. Women will be randomized 1:1 to GFA or Myomectomy (laparoscopic or abdominal).
  Interventions: Procedure: Global Fibroid Ablation (GFA); Procedure: Abdominal or Laparoscopic Myomectomy
- Woman Suitable for UAE or GFA (Active Comparator): This group will consist of women who desire uterine preservation. Women will be randomized 1:1 to GFA or uterine artery embolization (UAE).
  Interventions: Procedure: Global Fibroid Ablation (GFA); Procedure: Uterine Artery Embolization (UAE)

INTERVENTIONS:
Procedure: Global Fibroid Ablation (GFA) — GFA is being used for the treatment of symptomatic uterine fibroids
  Other Names: GFA
Procedure: Abdominal or Laparoscopic Myomectomy — Myomectomy is a procedure in which uterine fibroids are surgically removed from the uterus.
  Other Names: Myomectomy
  Arms: Woman Suitable for Myomectomy or GFA
Procedure: Uterine Artery Embolization (UAE) — UAE is a minimally invasive surgical procedure used to treat uterine fibroids.
  Other Names: UAE
  Arms: Woman Suitable for UAE or GFA

SUMMARY:
This Post Market study is being conducted to compare the direct and indirect cost of three approaches (GFA, myomectomy, and uterine artery embolization) for the treatment of symptomatic uterine fibroids.

DETAILED DESCRIPTION:
Uterine fibroids are the most common pelvic neoplasms in women; they severely impact quality of life and are the leading indication for hysterectomy. Hysterectomy is the definitive treatment for myomas; however, many patients seek alternative uterine-sparing therapy and desire to conserve their fertility. Myomectomy is a much-reported surgical option for women with symptomatic fibroids and, until recently, the abdominal approach has been the approach of choice for most surgeons. Over time, patients have requested less invasive procedures and minimally invasive, laparoscopic options are becoming more popular among patients and their gynecologists. Standard surgical and interventional treatments for uterine fibroids are costly to society and to the health care system. New technologies such as GFA may offer a low-cost alternative to the standard treatments for symptomatic uterine fibroids in women who desire uterine conservation. This study seeks to evaluate those cost differences between three available uterine-sparing techniques and to explore the qualitative outcomes such as symptom severity, health related quality of life, and overall treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years old and menstruating
* Have symptomatic uterine fibroids
* Have a uterine size ≤ 16 gestational weeks as determined by pelvic exam
* Have all fibroids that are less than 10 cm in any diameter
* Desire uterine conservation
* Have had a normal Pap smear within the past 36 months defined as "no untreated cervical malignancy or dysplasia."
* Are willing and able to comply with all study tests, procedures, and assessment tools
* Are capable of providing informed consent.

Exclusion Criteria:

* Have contraindications for laparoscopic surgery and/or general anesthesia.
* Are expected to be high risk for, or are known to have, significant intra-abdominal adhesions (defined as adhesions that would require extensive dissection to mobilize and view all surfaces of the uterus)
* Patients requiring major elective concomitant procedures (e.g., hernia repair)
* Are pregnant or lactating
* Have taken any depot GnRh agonist within three months prior to the screening procedures
* Have an implanted intrauterine or fallopian tube device for contraception that cannot or will not be removed at least 10 days prior to treatment
* Have chronic pelvic pain known to not be due to uterine fibroids
* Have known or suspected endometriosis Stage 3 or 4, adenomyosis
* Have active or history of pelvic inflammatory disease
* Have a history of, or evidence of, gynecologic malignancy or pre-malignancy within the past five years
* Have had pelvic radiation
* Have a non-uterine pelvic mass over 3 cm
* Have a cervical myoma
* Have one or more completely intracavitary submucous fibroids (Type 0) or only Type 0/1 submucous fibroids that are better treated via hysteroscopic methods
* In the medical judgment of the investigator should not participate in the study
* Are not willing to be randomized to treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-12; Primary Completion 2017-09 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Compare direct cost of GFA compared to those of myomectomy and UAE | 3 months post procedure
  To compare medical, surgical, and hospitalization costs (including procedural complication costs) of Global Fibroid Ablation (GFA) compared to those of Myomectomy and Uterine Artery Embolization (UAE)at 3 months post procedure.
Compare rates of acute and near-term serious complications to the acute and near-term treatment-related serious adverse events of pivotal study. | 3 months post procedure
  Overall rates of acute (within 48 hours post procedure) and near-term (between 2 and 30 days post procedure) serious complications in all GFA subjects compared to the acute and near-term treatment-related serious adverse event rates in the pivotal study.

SECONDARY OUTCOMES:
Assess the comparative safety of the three treatment alternatives | 60 Months
  Safety measures will be assessed by comparing the complication rate for all three alternatives (GFA, Myomectomy, UAE).
Assess factors that influence indirect costs of the three treatment alternatives | 60 Months
  Compare incidence costs of post discharge procedure-related complications and re-interventions we well as indirect cost factors defined as days to return-to-work, return to normal activities of daily living, and cost of care up to 60 months post discharge.
Assess UFS-QoL pre-treatment to post treatment in all treatment groups | 60 Months
  To compare fibroid symptom severity and quality of life scores at 3, 6, 12, 24, 36, 48, and 60 months post procedure as compared to baseline using the Uterine Fibroid Symptom and Health Related Quality of Life (UFS-QoL0 assessment tool.
Assess subjects menstrual bleeding using the MIQ | 60 Months
  Compare subjects menstrual bleeding pre-treatment and up to 3, 6, 12, 24, 36, 48, and 60 months post treatment using the Menorrhagia Impact Questionnaire (MIQ).
Assess subject's satisfaction with her treatment | 60 Months
  Compare subject's satisfaction and general health outcome at 3, 6, 12, 24, 36, 48, and 60 months post procedure as compared to baseline using the EQ-5D (a standardized instrument for use as a measure of health outcome).

CONTACTS AND LOCATIONS:
Overall Officials: John Thiel, MD, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (1):
- University of Saskatchewan, Saskatoon City Hospital, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Viswanathan M, Hartmann K, McKoy N, Stuart G, Rankins N, Thieda P, Lux LJ, Lohr KN. Management of uterine fibroids: an update of the evidence. Evid Rep Technol Assess (Full Rep). 2007 Jul;(154):1-122. PMID 18288885
- [Background] Twijnstra AR, Kolkman W, Trimbos-Kemper GC, Jansen FW. Implementation of advanced laparoscopic surgery in gynecology: national overview of trends. J Minim Invasive Gynecol. 2010 Jul-Aug;17(4):487-92. doi: 10.1016/j.jmig.2010.03.010. Epub 2010 May 14. PMID 20471917
- [Background] Holzer A, Jirecek ST, Illievich UM, Huber J, Wenzl RJ. Laparoscopic versus open myomectomy: a double-blind study to evaluate postoperative pain. Anesth Analg. 2006 May;102(5):1480-4. doi: 10.1213/01.ane.0000204321.85599.0d. PMID 16632830
- [Background] Parker WH, Iacampo K, Long T. Uterine rupture after laparoscopic removal of a pedunculated myoma. J Minim Invasive Gynecol. 2007 May-Jun;14(3):362-4. doi: 10.1016/j.jmig.2006.10.024. PMID 17478371
- [Background] Banas T, Klimek M, Fugiel A, Skotniczny K. Spontaneous uterine rupture at 35 weeks' gestation, 3 years after laparoscopic myomectomy, without signs of fetal distress. J Obstet Gynaecol Res. 2005 Dec;31(6):527-30. doi: 10.1111/j.1447-0756.2005.00331.x. PMID 16343253
- [Background] Moss JG, Cooper KG, Khaund A, Murray LS, Murray GD, Wu O, Craig LE, Lumsden MA. Randomised comparison of uterine artery embolisation (UAE) with surgical treatment in patients with symptomatic uterine fibroids (REST trial): 5-year results. BJOG. 2011 Jul;118(8):936-44. doi: 10.1111/j.1471-0528.2011.02952.x. Epub 2011 Apr 12. PMID 21481151
- [Background] Mara M, Maskova J, Fucikova Z, Kuzel D, Belsan T, Sosna O. Midterm clinical and first reproductive results of a randomized controlled trial comparing uterine fibroid embolization and myomectomy. Cardiovasc Intervent Radiol. 2008 Jan-Feb;31(1):73-85. doi: 10.1007/s00270-007-9195-2. Epub 2007 Oct 18. PMID 17943348
- [Background] Manyonda IT, Bratby M, Horst JS, Banu N, Gorti M, Belli AM. Uterine artery embolization versus myomectomy: impact on quality of life--results of the FUME (Fibroids of the Uterus: Myomectomy versus Embolization) Trial. Cardiovasc Intervent Radiol. 2012 Jun;35(3):530-6. doi: 10.1007/s00270-011-0228-5. Epub 2011 Jul 20. PMID 21773858
- [Background] Carls GS, Lee DW, Ozminkowski RJ, Wang S, Gibson TB, Stewart E. What are the total costs of surgical treatment for uterine fibroids? J Womens Health (Larchmt). 2008 Sep;17(7):1119-32. doi: 10.1089/jwh.2008.0456. PMID 18687032
- [Background] Nash K, Feinglass J, Zei C, Lu G, Mengesha B, Lewicky-Gaupp C, Lin A. Robotic-assisted laparoscopic myomectomy versus abdominal myomectomy: a comparative analysis of surgical outcomes and costs. Arch Gynecol Obstet. 2012 Feb;285(2):435-40. doi: 10.1007/s00404-011-1999-2. Epub 2011 Jul 22. PMID 21779774
- [Background] Al-Fozan H, Dufort J, Kaplow M, Valenti D, Tulandi T. Cost analysis of myomectomy, hysterectomy, and uterine artery embolization. Am J Obstet Gynecol. 2002 Nov;187(5):1401-4. doi: 10.1067/mob.2002.127374. PMID 12439538
- [Background] Bushnell DM, Martin ML, Moore KA, Richter HE, Rubin A, Patrick DL. Menorrhagia Impact Questionnaire: assessing the influence of heavy menstrual bleeding on quality of life. Curr Med Res Opin. 2010 Dec;26(12):2745-55. doi: 10.1185/03007995.2010.532200. Epub 2010 Nov 3. PMID 21043553
- [Background] Hartung J, Knapp G. On tests of the overall treatment effect in meta-analysis with normally distributed responses. Stat Med. 2001 Jun 30;20(12):1771-82. doi: 10.1002/sim.791. PMID 11406840
- [Background] Chudnoff SG, Berman JM, Levine DJ, Harris M, Guido RS, Banks E. Outpatient procedure for the treatment and relief of symptomatic uterine myomas. Obstet Gynecol. 2013 May;121(5):1075-1082. doi: 10.1097/AOG.0b013e31828b7962. PMID 23635746
- [Background] Robles R, Aguirre VA, Argueta AI, Guerrero MR. Laparoscopic radiofrequency volumetric thermal ablation of uterine myomas with 12 months of follow-up. Int J Gynaecol Obstet. 2013 Jan;120(1):65-9. doi: 10.1016/j.ijgo.2012.07.023. Epub 2012 Oct 14. PMID 23073229
- [Background] Garza Leal JG, Hernandez Leon I, Castillo Saenz L, Lee BB. Laparoscopic ultrasound-guided radiofrequency volumetric thermal ablation of symptomatic uterine leiomyomas: feasibility study using the Halt 2000 Ablation System. J Minim Invasive Gynecol. 2011 May-Jun;18(3):364-71. doi: 10.1016/j.jmig.2011.02.006. PMID 21545960
- [Background] Guido RS, Macer JA, Abbott K, Falls JL, Tilley IB, Chudnoff SG. Radiofrequency volumetric thermal ablation of fibroids: a prospective, clinical analysis of two years' outcome from the Halt trial. Health Qual Life Outcomes. 2013 Aug 13;11:139. doi: 10.1186/1477-7525-11-139. PMID 23941588
- [Background] Macer JA. For uterine-sparing fibroid treatment, consider laparoscopic ultrasound-guided radiofrequency ablation. obmanagement.com Vol 25 No. 11 November 2013
- [Background] Berman JM, Guido RS, Garza Leal JG, Pemueller RR, Whaley FS, Chudnoff SG; Halt Study Group. Three-year outcome of the Halt trial: a prospective analysis of radiofrequency volumetric thermal ablation of myomas. J Minim Invasive Gynecol. 2014 Sep-Oct;21(5):767-74. doi: 10.1016/j.jmig.2014.02.015. Epub 2014 Mar 5. PMID 24613404